CLINICAL TRIAL: NCT06918691
Title: The Effect Of Technology Addiction Prevention Program On University Students At Risk For Technology Addiction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Çiçek Önder, M.Sc., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IUC-NURSE-CO-01
Record Dates: First submitted 2025-03-17; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Technology Addiction; Public Health Nursing; School Health
Keywords: school health; public health nursing; technology addiction
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- education (Experimental): The group that received a 7-week technology addiction prevention program
  Interventions: Behavioral: technology addiction prevention program
- plasebo (No Intervention): The group that received a 7-week technology addiction prevention program

INTERVENTIONS:
Behavioral: technology addiction prevention program — technology addiction prevention program
  Arms: education

SUMMARY:
Due to the increasing use of technological devices among adolescents, technology addiction is a serious public health problem that requires intervention. In order to cope with this problem, it is necessary to develop programs that have proven effects and are suitable for our culture and the psychosocial development of the age group in question. In the project planned to be carried out in two stages, university students at risk of technology addiction will be identified and the effect of the developed technology addiction prevention program will be evaluated. In these days when national combat studies on behavioral addictions are initiated in our country, the results of the research will contribute to the development of national action plans in the fight against technology addiction. The purpose of this doctoral thesis is to evaluate the effect of the technology addiction prevention program for university students at risk of technology addiction.

DETAILED DESCRIPTION:
Although it is generally used for leisure purposes, the increase in technological device and internet use affects all age groups and has positive and negative effects on public health. These effects lead to various behavioral problems, especially in adolescents. As a result of the unconscious, excessive, uncontrolled and pathological use of technological devices, behavioral mental health problems such as "technology addiction" emerge. When some studies revealing the prevalence of game addiction among adolescents in European countries are examined, it is seen that it varies between 2.2% and 30.4%. In studies in Türkiye, according to the results of the research conducted by the Turkish Statistical Institute (TÜİK) with children aged 6-15 in 2021, internet usage rates in children were 82.7% and regular internet usage rates increased. It was found that internet usage and gaming rates were higher in boys than in girls. It is seen that the purpose of internet use is first for homework or learning purposes with 84.8% and second for playing games with 79.5%. 31.3% of children who use the internet regularly used social media. According to TUİK 2013 data, the rate of children who own at least one information technology product has increased. Many physical and psychological changes are observed during adolescence. Individuals' lifestyles and healthy life behaviors are shaped during this period. It is accepted that the use of technological tools and equipment, internet use and moderate gaming as part of a healthy lifestyle can have many positive effects such as emotional relaxation, strong peer support and social bonding. Behavioral problems arise as a result of excessive and uncontrolled use of technological tools. The main health problems that arise due to problematic technological tool and equipment use behavior include inadequate physical activity, unhealthy nutrition, vision or hearing problems, musculoskeletal system problems, sleep disorders, psychological problems such as depression, venous health problems such as thromboembolism and decreased academic success. Model-based approaches are needed to prevent health problems that arise in individuals as a result of problematic health behaviors and to create and develop positive healthy behaviors. Therefore, in this study, an educational program will be created using Cox's Health Behavior Interaction Model (SDEM) as a conceptual framework to evaluate the variables that affect university students' problematic technology use behaviors, the relationships between these variables, and to gain positive health behaviors. This study aims to evaluate the effect of a technology addiction prevention program for university students at risk of technology addiction.

ELIGIBILITY:
Inclusion Criteria:

* University students who scored 37 and above on the young internet addiction test short form
* University students who scored 49 and above on the technology addiction scale
* First grade university students

Exclusion Criteria:

* Mentally unstable

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
young internet addiction test short form | Baseline, Immediately after post-test, month 3 after the post test, month 6 after the post test
  The internet addiction levels of university students will be determined with the technology addiction prevention program.
technology addiction scale | Baseline, Immediately after post-test, month 3 after the post test, month 6 after the post test
  The technology addiction levels of university students will be determined with the technology addiction prevention program.
screen time | Baseline, Immediately after post-test, month 3 after the post test, month 6 after the post test
  It will be used to measure students' screen time before the test, after the test and during follow-up.
number of steps | Baseline, Immediately after post-test, month 3 after the post test, month 6 after the post test
  Raising awareness to increase physical activity through a technology addiction prevention program

SECONDARY OUTCOMES:
sleeping duration | Baseline, Immediately after post-test, month 3 after the post test, month 6 after the post test
  It will be determined whether there is any change in the student during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Çiçek ÖNDER, Principal Investigator — Istanbul University - Cerrahpasa; Aysun ARDIÇ, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Beykent University, Istanbul, BEYLİKDÜZÜ., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want it to be visible

REFERENCES:
- See also: World health organization — https://www.who.int/europe/news/item/25-09-2024-teens--screens-and-mental-health